CLINICAL TRIAL: NCT06183333
Title: Efficacy of a Web-Based Emotion Regulation Training in a Transdiagnostic Sample: A Randomized Controlled Trial
Brief Title: Efficacy of a Web-Based Emotion Regulation Training in a Transdiagnostic Sample
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Luise Pruessner, Principal Investigator, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ER-Training
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Emotion Regulation; Anxiety Disorders; Depression; Eating Disorders; Borderline Personality Disorder
Keywords: Internet-Based Intervention; Web-Based Training; Emotion Regulation
MeSH Terms: conditions — Emotional Regulation; Anxiety Disorders; Depression; Feeding and Eating Disorders; Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with an Intervention Group and a Waiting List Control Group
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical interviews and data analysis will be conducted blindly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Web-based emotion regulation intervention
  Interventions: Behavioral: Heidelberg Emotion Regulation Training
- Waitlist control group (No Intervention): Eight-week waiting period

INTERVENTIONS:
Behavioral: Heidelberg Emotion Regulation Training — The four-week intervention program is specifically designed to enhance the participants' emotion regulation. It focuses on developing their skills in accurately recognizing various emotions and effectively applying diverse emotion regulation strategies. To achieve this, the program includes video-based psychoeducation sessions. Alongside these sessions, the program incorporates daily short exercises, each lasting approximately five minutes. These exercises are crafted to help participants practically integrate the concepts and strategies learned from the psychoeducation sessions into their everyday lives. All components of the intervention are accessible through an online platform, ensuring ease of access and flexibility for participants.
  Arms: Intervention group

SUMMARY:
This two-armed randomized controlled trial investigates the efficacy of a web-based emotion regulation intervention in a transdiagnostic sample. The sample includes participants diagnosed with anxiety disorders, depression, eating disorders, borderline personality disorder, and healthy controls without a current psychiatric diagnosis. Participants will be randomly assigned to either the intervention group, receiving a web-based emotion regulation program, or a waitlist control group, which will have delayed intervention access after eight weeks.

The intervention is grounded in cognitive-behavioral therapy (CBT), featuring everyday emotion regulation exercises, and psychoeducation delivered through video and audio files. Outcome measures include emotion regulation abilities, well-being, anxiety, depression, eating disorder symptoms, personality pathology, and self-esteem, evaluated at four and eight weeks post-baseline.

DETAILED DESCRIPTION:
Background:

Emotion regulation is pivotal in the pathogenesis and persistence of diverse psychopathologies. While anxiety disorders are often marked by an impaired ability to modulate acute fear responses, depressive disorders feature enduring negative affect and frequent rumination. In eating disorders, emotional dysregulation typically leads to maladaptive coping via disordered eating behaviors, whereas in borderline personality disorder, it manifests as emotional instability. The pervasiveness of emotion regulation difficulties across these diverse clinical presentations highlights a need for treatments targeting this shared mechanism. Our study aims to address this gap by testing the effectiveness of a novel web-based emotion regulation intervention in a transdiagnostic sample.

Method:

This two-armed randomized controlled trial involves participants aged 18 and above diagnosed with anxiety disorders, depression, eating disorders, borderline personality disorder, and healthy controls without psychiatric diagnoses. Participants will be randomly assigned to one of two groups:

1. Web-based emotion regulation intervention.
2. Waitlist control group with delayed intervention access (eight weeks).

The intervention, accessible via mobile phones or desktop browsers, employs cognitive-behavioral therapy (CBT) techniques, offering everyday emotion regulation exercises and psychoeducation through video material and audio files.

Outcome measures, including emotion regulation abilities, well-being, anxiety, depression, eating disorder symptoms, personality pathology, and self-esteem, will be assessed at four and eight weeks post-baseline.

Hypotheses:

The intervention is expected to result in improved emotion regulation abilities and well-being, along with reduced anxiety, depression, eating disorder symptoms, personality pathology, and self-esteem compared to the waitlist control group. The transdiagnostic intervention is anticipated to demonstrate superiority in addressing the diverse emotional challenges across different psychological disorders.

Additional Laboratory Study:

A subgroup of participants will be invited for a follow-up laboratory assessment of physiological indicators of emotion regulation abilities four weeks after their initial baseline measurement. We hypothesize that the intervention will lead to notable improvements in implicit emotion regulation capacity measured during a resting period and the presentation of negative emotional images. Furthermore, we anticipate observable improvements in explicit emotion regulatory skills, specifically in the downregulation of negative emotions and the upregulation of positive emotions, as assessed through a picture-viewing paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient German language skills (C1)
* Permanent internet access during the study period
* ≥ 18 years of age

Exclusion Criteria:

* Acute suicidality
* Current severe substance use disorder
* Current severe depressive episode
* Lifetime bipolar disorder
* Lifetime psychotic disorders
* Body Mass Index (BMI) below 18.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Emotion Regulation Difficulties | 0 weeks, 4 weeks, 8 weeks
  The Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004)

SECONDARY OUTCOMES:
Changes in Emotion Regulation Strategy Use | 0 weeks, 4 weeks, 8 weeks
  The Heidelberg Form for Emotion Regulation Strategies (HFERST; Izadpanah et al., 2019)
Changes in Well-Being | 0 weeks, 4 weeks, 8 weeks
  The World Health Organization Well-Being Index (WHO-5; Topp et al., 2015)
Changes in Anxiety Symptoms | 0 weeks, 4 weeks, 8 weeks
  The General Anxiety Disorder Scale (GAD-7; Spitzer et al., 2006)
Changes in Depressive Symptoms | 0 weeks, 4 weeks, 8 weeks
  The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001)
Changes in Eating Psychopathology | 0 weeks, 4 weeks, 8 weeks
  The Eating Disorders Examination Questionnaire (EDE-Q; Berg et al., 2012)
Changes in Personality Pathology | 0 weeks, 4 weeks, 8 weeks
  The Personality Inventory for DSM-5 (PID-5; Krueger et al., 2012)
Changes in Eating-Disorder-Related Daily Difficulties | 0 weeks, 4 weeks, 8 weeks
  The Clinical Impairment Assessment Questionnaire (CIA; Bohn et al., 2008)
Changes in Self-Esteem | 0 weeks, 4 weeks, 8 weeks
  The Rosenberg Self-Esteem Scale (RSES; Roth et al., 2008)
Changes in Weekly Emotion Regulation Strategy Use | 0 weeks, 1 weeks, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks
  Weekly assessment of emotion regulation strategies (adapted from Pruessner et al., 2023).
Changes in Weekly Positive and Negative Affect | 0 weeks, 1 weeks, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks
  Positive and Negative Affect Schedule - Expanded Form (16 items; PANAS-X; Watson & Clark, 1994)
Changes in Weekly Eating Psychopathology | 0 weeks, 1 weeks, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks
  The Eating Disorders Examination Questionnaire (EDE-QS; Gideon et al., 2016)

OTHER OUTCOMES:
Implicit Emotion Regulation Capacity | 4 weeks
  Responses to negative images (corrugator electromyogram, frontal alpha asymmetry, affect ratings) and heart rate variability during a laboratory resting period (Thayer & Lane, 2000)
Negative Emotion Downregulation Ability | 4 weeks
  Changes in responses to negative images (corrugator electromyogram, frontal alpha asymmetry, affect ratings) following a downregulation instruction in a laboratory emotion regulation task (adapted from Ertl et al., 2013)
Positive Emotion Upregulation Ability | 4 weeks
  Changes in responses to positive images (corrugator electromyogram, frontal alpha asymmetry, affect ratings) following an upregulation instruction in a laboratory emotion regulation task (adapted from Cheng et al., 2023)

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Hartmann, Principal Investigator — Department of Psychology, Heidelberg University; Luise Pruessner, Principal Investigator — Department of Psychology, Heidelberg University; Sven Barnow, PhD, Study Chair — Department of Psychology, Heidelberg University; Daniel V. Holt, PhD, Study Chair — Department of Psychology, Heidelberg University
Locations (1):
- Heidelberg University, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available after the publication of the study results.
Access Criteria: Open access, available upon request to ensure appropriate use.
URL: http://osf.io

REFERENCES:
- [Background] Ritschel LA, Tone EB, Schoemann AM, Lim NE. Psychometric properties of the Difficulties in Emotion Regulation Scale across demographic groups. Psychol Assess. 2015 Sep;27(3):944-54. doi: 10.1037/pas0000099. Epub 2015 Mar 16. PMID 25774638
- [Background] Izadpanah S, Barnow S, Neubauer AB, Holl J. Development and Validation of the Heidelberg Form for Emotion Regulation Strategies (HFERST): Factor Structure, Reliability, and Validity. Assessment. 2019 Jul;26(5):880-906. doi: 10.1177/1073191117720283. Epub 2017 Jul 21. PMID 28730850
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Hilbert A, de Zwaan M, Braehler E. How frequent are eating disturbances in the population? Norms of the eating disorder examination-questionnaire. PLoS One. 2012;7(1):e29125. doi: 10.1371/journal.pone.0029125. Epub 2012 Jan 18. PMID 22279527
- [Background] Zimmermann J, Altenstein D, Krieger T, Holtforth MG, Pretsch J, Alexopoulos J, Spitzer C, Benecke C, Krueger RF, Markon KE, Leising D. The structure and correlates of self-reported DSM-5 maladaptive personality traits: findings from two German-speaking samples. J Pers Disord. 2014 Aug;28(4):518-40. doi: 10.1521/pedi_2014_28_130. Epub 2014 Feb 10. PMID 24511899
- [Background] Roth M, Altmann T. A Comparison of the Predictive Validity of Self-Esteem Level and Directly Measured Self-Esteem Stability in the Temporal Prediction of Psychological Distress. Front Psychol. 2020 Jul 24;11:1770. doi: 10.3389/fpsyg.2020.01770. eCollection 2020. PMID 32849049